CLINICAL TRIAL: NCT03749759
Title: Pain Perception and Discomfort of Second Eye Cataract Surgery in Comparison With the First Eye in Correlation With Perioperative Stress
Brief Title: Perioperative Stress and Pain Perception of Second Eye Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Neuromaster
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; Biofeedback
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biofeedback measurement (Experimental): A Biofeedback measurement will be done during cataract surgery of both eyes
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — A biofeedback measurement will be carried out during cataract surgery of both eyes

SUMMARY:
Purpose of this study is to find a correlation between agitation (stress) indicating parameters and the pain perception during second eye cataract surgery, compared to first eye cataract surgery.

DETAILED DESCRIPTION:
A cataract, which is the clouding of the eye's natural lens as a result of aging or injury, is the leading cause of preventable blindness worldwide. As one of the of the most common surgical procedures, cataract surgery is performed almost 22 million times worldwide each year. The World Health Organisation estimates that by 2020 more than 32 million cataract surgeries will take place globally per annum.

Phacoemulsification cataract surgery in topical anaesthesia has become the anaesthetic method of choice since first described by Fichman in 1992. Although this procedure has proven to be relatively painless, safe and effective, patients often report increased pain or discomfort during surgery of the second eye. Several studies were performed to find out if there was any proof to that common finding and some tried to find a correlation to fear and anxiety using standardized questionnaires.

In one study of 65 patients there was a subtle increase in pain in the second surgery relative to the first which appeared to be associated with decreased preoperative anxiety. Another study found that previous cataract extraction correlated negatively, but weakly with preoperative anxiety.

A study of 70 patients having first cataract extraction found no difference in mean pain scores, fear and anxiety when compared with a second, independent population of 57 patients having second cataract extraction. A similar outcome was found in 2 other studies where there was no difference in perceived pain between the first and second cataract surgery.

Summarized, the results in the related literature are controversial concerning the assessment of pain, fear and anxiety during cataract surgery performed in the second eye.

Emotional stress and anxiety in surgical patients lead to sympathetic stimulation with tachycardia, hypertension and possible cardiac ischaemia which are haemodynamic stress responses, triggered by endocrine regulatory mechanisms and the autonomic nervous system with increased cortisol, adrenaline and noradrenaline blood levels. Furthermore palmar and plantar sweat glands activity decreases skin resistance which is shown as a surge in electric skin conductance in bio- feedback measurements.

For obtaining and processing the information about these physiological reactions a system with the ability to measure and record various bio-signals is needed. These kind of systems are used for biofeedback. Galvanic Skin response Sensors measure the above mentioned electrical conductance of the skin. It is used as an indication of psychological and physiological excitation and thus represents an indicator for the individual's stress response.

Electromyograph (EMG) uses surface electrodes to measure the electrical activity of the skeletal muscles when they are relaxed and contracted by detecting the combined electrical potential generated by the muscle cells. The mean value of the rectified EMG signal of the upper trapezius muscle increases during stressful conditions and decreases again during relaxation periods.

Electrocardiogram (ECG) electrodes are used to measure the heart function and further calculate the heart rate variability (HRV). HRV is defined as the beat-to-beat changes, the interbeat interval, which is the time between two successive R waves. HRV is considered as a measure of the interaction between sympathetic and parasympathetic influence on heart rate. The activation of the sympathetic branch of the autonomic nervous system increases heart rate, while the activation of the parasympathetic branch, primarily mediated by the vagus nerve, slows it. These physiological signals provide a reliable measurement of agitation (stress).

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* written informed consent prior to surgery
* bilateral age-related cataract

Exclusion Criteria:

* deafness
* allergy to topical anesthetic agents
* severe anxiety and involuntary eye and head movements
* conditions likely to require surgical therapy other than routine phacoemulsification (eg: traumatic and complicated cataracts)
* in case of pregnancy (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative agitation (stress) measurement | 12 months
  Perioperative stress will be measured using the BioLink Biofeedback device, which records an electrocardiogram, an electromyogram, skin conductance and respiratory rate. Changes in the different values show how stressed the patient was during the surgeries.

SECONDARY OUTCOMES:
Assessment of pain perception | 12 months
  Pain perception of the patients will be assessed during the two cataract surgeries using an visual analogue scale, where 10 means highest pain and 1 is lowest pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided